CLINICAL TRIAL: NCT05150613
Title: Individual Performance Analysis of Cardiopulmonary Exercise Testing / Maximal and Sub-maximal Exercise Testing With Different Face Masks
Brief Title: Impact of Different Face Masks on Maximal and Submaximal Performance Testing During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Syeda Rida Batool
Record Dates: First submitted 2021-11-23; First posted 2021-12-09 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
Keywords: Face masks; COVID-19; Maximal Test; Submaximal Test; Surgical mask; N95 mask
MeSH Terms: conditions — COVID-19 | interventions — N95 Respirators

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinding method will be employed to limit possible participant influence on test results (anticipation bias)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Other): No Mask
  Interventions: Other: No Mask; Other: Surgical Mask; Other: N95 Mask
- Group B (Other): Surgical Mask
  Interventions: Other: No Mask; Other: Surgical Mask; Other: N95 Mask
- Group C (Other): N95 Mask
  Interventions: Other: No Mask; Other: Surgical Mask; Other: N95 Mask

INTERVENTIONS:
Other: No Mask — Participants fulfilling inclusion exclusion criteria will be asked to sign informed consent. Sealed envelope randomization method would determine order of testing (Group A; No mask, Group B; Surgical mask, Group C; N95 mask). For 6MWT, participants will be asked to walk on 30-meter unimpeded walkway as much as possible & distance at end is recorded along with number of stops during test. For Bruce Protocol, participants will follow standard stage succession with an abrupt increase in speed & inclination by end of each 3-minute cycle. The participants will be advised to perform test till exhaustion and level achieved will be recorded. The analyzed data will then be used to calculate VO2max and MET scores. Heart rate, SPO2, respiratory rate will be recorded at baseline, after 2 minutes and at test completion. BP will be recorded at baseline and at completion of test, while perceived discomfort scale & post-exercise exhaustion scale will be assessed upon completion of exercise testing.
Other: Surgical Mask — Participants fulfilling inclusion exclusion criteria will be asked to sign informed consent. Sealed envelope randomization method would determine order of testing (Group A; No mask, Group B; Surgical mask, Group C; N95 mask). For 6MWT, participants will be asked to walk on 30-meter unimpeded walkway as much as possible & distance at end is recorded along with number of stops during test. For Bruce Protocol, participants will follow standard stage succession with an abrupt increase in speed & inclination by end of each 3-minute cycle. The participants will be advised to perform test till exhaustion and level achieved will be recorded. The analyzed data will then be used to calculate VO2max and MET scores. Heart rate, SPO2, respiratory rate will be recorded at baseline, after 2 minutes and at test completion. BP will be recorded at baseline and at completion of test, while perceived discomfort scale & post-exercise exhaustion scale will be assessed upon completion of exercise testing.
Other: N95 Mask — Participants fulfilling inclusion exclusion criteria will be asked to sign informed consent. Sealed envelope randomization method would determine order of testing (Group A; No mask, Group B; Surgical mask, Group C; N95 mask). For 6MWT, participants will be asked to walk on 30-meter unimpeded walkway as much as possible & distance at end is recorded along with number of stops during test. For Bruce Protocol, participants will follow standard stage succession with an abrupt increase in speed & inclination by end of each 3-minute cycle. The participants will be advised to perform test till exhaustion and level achieved will be recorded. The analyzed data will then be used to calculate VO2max and MET scores. Heart rate, SPO2, respiratory rate will be recorded at baseline, after 2 minutes and at test completion. BP will be recorded at baseline and at completion of test, while perceived discomfort scale & post-exercise exhaustion scale will be assessed upon completion of exercise testing.

SUMMARY:
In COVID 19, masks wearability has become a new normal and this "new normal" presented evidence-based performance limitations. The study findings are aimed to objectify parametric changes (if any) and therefore, will assist in making future decisions for testing programs with minimum limitation and maximum protection in this pandemic.

DETAILED DESCRIPTION:
Victimizing millions of individuals, the novel coronavirus (COVID-19) has made drastic changes in our lives including the obligation of personal protective equipment (PPEs), especially masks. This obligation presented evidence-based performance limitations owing to mask associated airflow resistance, increased ventilatory effort, external air trapping thus elevated carbon dioxide concentration and reuptake, thermal effects, and ventilatory parameters decline along with other physiological, psychological and health-related consequences.

Despite the reported success of vaccination, the use of PPEs especially face masks as one of the non-pharmacological solution to limit viral transmission is a controversial recommendation. With diameter difference between SARS-CoV-2 and mask threads makes viral transmission non-preventable, it however could be reduced partially from 67% to 17% due to the filtration barrier provided by face masks. With new research supporting viral transmission from asymptomatic individuals, the United States Centre of Disease Control (CDC) recommends the use of face masks in an indoor and outdoor setting requiring public interaction where social distancing is unrealistic.

Cardio Pulmonary Exercise Testing (CPET) is an important clinical tool to assess aerobic capacity and has value in predicting outcomes not only in cardiac diseased populations but in other conditions also. Being a gold standard for risk stratification and exercise prescription plans, its application sometimes becomes impractical and thus formulation and utilization of submaximal and graded exercises test proved fruitful in rehabilitation program design in terms of cost efficiency and little expertise requirement for performance. With pandemic in place, the procedure for exercise testing has changed from routine practice. The addition of masks during testing procedures, as per recommendations of CDC to avoid cross-contamination among the health care providers and the participating community, as aerosol generation during exercise testing as a consequence of frequent forceful respiration due to variable exercise intensities thus high discharge rates and farther viral spread.

Both submaximal (6MWT) and maximal (Bruce protocol) exercise tests are commonly used exercise tests in a health care setting with high prognostic and diagnostic values. As per knowledge, there is limited evidence available on testing procedure and therefore the plan is to cover the gaps identified in previous research based on 6MWT and Bruce protocol (mask variability, sample modesty, age restrictions; data on young healthy individuals, few analyzed testing parameters) and note the performance differences if achieved to guide the formulation of structured and standardized approach towards both testing procedures using medically acceptable masks as a general requirement for future testing. As no guidelines had yet been issued to adapt the testing to current situations with PPEs. Analysis of parametric changes in healthy volunteers would aid in the formulation of a recommendation plan for performance analysis measures used in cardiopulmonary settings to ensure minimum performance limitation with added equipment and maintenance of consistency in adaptive testing.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Population from all age groups
* Healthy Individuals
* Physically active - screening through Get Active questionnaire
* Willing to consent

Exclusion Criteria:

* Cognitively Impaired
* Participants with absolute or relative contraindication to exercise testing
* Underlying condition limiting mask wearability
* Communication gap (language other than Urdu or English)
* Subjects performing regular physical activity (sports personal)
* Latent known/diagnosed disease condition
* People with Long Covid (evaluated via self-reported Post COVID-19 Functional Status Scale)
* Patients with laboratory diagnosed and symptomatic COVID-19

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
6MWT (Marked Walking Course, Stop Watch) | After 48 hours
  6mwt is a submaximal testing procedure developed by the American Thoracic Society to assess aerobic capacity, endurance, and changes in performance capacity. The test measures the distance covered in 6 Minutes and is intended for all populations with a wide range of diagnoses. The procedure requires a 30-meter unimpeded walkway, a timer, distance markers, turning pointers (cones) and monitoring gadgets (oximeter, Borg's scale), and chairs for the resting period (on requirement). The participants are instructed to walk as much as possible with minimum rests and regular standardized encouragements are provided throughout the test. The distance at the end is recorded along with the number of stops during the test and other parameters. Low distance scores are indicative of reduced performance capacity.
  It will be used for sub maximal testing of participants with no mask, surgical mask and wearing N95 mask with the minimum wash out period of 48 hours.
Bruce Protocol (Treadmill) | After 48 hours
  The standard Bruce protocol is the most preferred exercise stress test with validated outcomes and good prognostic values. It is a standard test in cardiology and is divided into successive stages of 3 minutes with an abrupt increase in speed and inclination by the end of each 3-minute cycle. Bruce protocol has 7 stages with starting speed of 1.7 miles/h at 10% inclination (2% inclination increase/stage). The speed change follows as; Level 2 (2.5 miles/h), level 3 (3.4 miles/h), level 4 (4.2 miles/h), level 5 (5.0 miles/h), level 6 (5.5 miles/h) and level 7 (6.0 miles/h) respectively. The participants are advised to perform the test till exhaustion, or the test is suspended based on unlikely events. It will be used for maximal testing of participants with no mask, surgical mask and wearing N95 mask with the minimum wash out period of 48 hours.

SECONDARY OUTCOMES:
Modified Borg's Scale for Rate of Perceived Exertion (RPE) (Dyspnea Score) | After 1minute
  Modified Borg's scale is a validated and reliable outcome measure to rate subjective perception of exertion and breathlessness. A commonly employed tool used in cardiopulmonary rehabilitation to monitor progress in rehabilitation programs. Borg's scale, the modified version of the original scale proposed by Gunner, is mostly used in the diagnosis of effort-related dyspnea, chest pain, and musculoskeletal pain. The scale consists of a grading score from 0-10 (0; being no exertion at all to 10; being maximal). Subjective perception is rated during the activity. The chosen number from the numeric list denotes the intensity of activity allowing to speed up or slow down activity. The scale takes a few seconds to record responses and can be administered single or multiple times during the process.
Discomfort Perception Scale | After 2 minutes
  The discomfort scale is utilized to rate subjective perception about ten sensations of discomfort (Humidity, heat, breathing resistance, itchiness, tightness, saltiness, feeling unfit, odor, fatigue, and overall discomfort). The scale has A 10-point rating scale for response record with 0 representing "none", 5 representing "acceptable" and 10 "very fond of." Low individual scores are indicative of low level of associated discomfort while high scores correspond to greater subjective discomfort perception.
Hecimovich-Peiffer-Harbaugh Exercise Exhaustion Scale | After 5minutes
  The post-exercise exhaustion scale is a validated and reliable tool to assess exercise-induced acute onset of exhaustion. The scale consists of 14 items that are measured by a 10-point Likert type frequency/intensity scale of response categories anchored at extreme ends by 'not at all to 'extremely difficult'. High scores are associated with elevated post-exercise exhaustion.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah Rehabilitation Center, Islamabad, AL
  - Riphah International University, Islamabad, Federal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egger F, Blumenauer D, Fischer P, Venhorst A, Kulenthiran S, Bewarder Y, Zimmer A, Bohm M, Meyer T, Mahfoud F. Effects of face masks on performance and cardiorespiratory response in well-trained athletes. Clin Res Cardiol. 2022 Mar;111(3):264-271. doi: 10.1007/s00392-021-01877-0. Epub 2021 Jun 6. PMID 34091726
- [Background] Shaw K, Butcher S, Ko J, Zello GA, Chilibeck PD. Wearing of Cloth or Disposable Surgical Face Masks has no Effect on Vigorous Exercise Performance in Healthy Individuals. Int J Environ Res Public Health. 2020 Nov 3;17(21):8110. doi: 10.3390/ijerph17218110. PMID 33153145
- [Background] Fikenzer S, Uhe T, Lavall D, Rudolph U, Falz R, Busse M, Hepp P, Laufs U. Effects of surgical and FFP2/N95 face masks on cardiopulmonary exercise capacity. Clin Res Cardiol. 2020 Dec;109(12):1522-1530. doi: 10.1007/s00392-020-01704-y. Epub 2020 Jul 6. PMID 32632523
- [Background] Lassing J, Falz R, Pokel C, Fikenzer S, Laufs U, Schulze A, Holldobler N, Rudrich P, Busse M. Effects of surgical face masks on cardiopulmonary parameters during steady state exercise. Sci Rep. 2020 Dec 21;10(1):22363. doi: 10.1038/s41598-020-78643-1. PMID 33349641
- [Background] Shein SL, Whitticar S, Mascho KK, Pace E, Speicher R, Deakins K. The effects of wearing facemasks on oxygenation and ventilation at rest and during physical activity. PLoS One. 2021 Feb 24;16(2):e0247414. doi: 10.1371/journal.pone.0247414. eCollection 2021. PMID 33626065
- [Background] Swiatek KM, Lester C, Ng N, Golia S, Pinson J, Grinnan D. Impact of Face Masks on 6-Minute Walk Test in Healthy Volunteers. Pulm Circ. 2021 Jan 20;11(1):2045894020988437. doi: 10.1177/2045894020988437. eCollection 2021 Jan-Mar. PMID 33532062